CLINICAL TRIAL: NCT01218243
Title: An Efficacy Trial of Electroacupuncture at Points of Bilateral BL33 for Mild and Moderate Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Dean of Acupuncture Department of Guangan'men Hospital, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009S208
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Acupuncture; Mild and moderate BPH
MeSH Terms: conditions — Prostatic Hyperplasia; Lymphoma, Follicular | interventions — Needles; Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acupoint (Experimental): Needle at bilateral BL33 60-80 mm with a 45°angle.A feeling of soreness and distension will be felt when needling into the 3rd posterior sacral foramina(S3).Needle with a 100-125 mm long needle without lifting, thrusting or rotating.G6805-2 electric stimulator (produced by Shanghai Huayi Medical Instrument Co.Ltd)is put on with Sparse-dense wave,20Hz. Stop turning up the current intensity when patients could not stand. There are 5 sessions in the first two weeks and 3 sessions in the last two weeks, 30 min/session.
  Interventions: Device: needle
- non-acupoint (Sham Comparator): Take the place 2 cun far from BL33 on the outside horizontally as the non-point. Needle on the non-point for 60-80mm with a 45°angle. A feeling of soreness and distension will be felt .Needle with a 100-125mm long needle without lifting, thrusting or rotating.Sparse-dense wave,20Hz. Stop turning up the current intensity when patients could not stand. 5 times for the first two weeks and 3 times for the last two weeks, 30 min/time.
  Interventions: Device: needle

INTERVENTIONS:
Device: needle — For the acupoint group,needle on bilateral BL33 60-80mm with a 45°angle. A feeling of soreness and distension will be felt when needling into the 3rd posterior sacral foramina(S3).Needle with a 100-125 mm long needle without lifting, thrusting or rotating.An electric stimulator is put on.G6805-2 electric stimulator (produced by Shanghai Huayi Medical Instrument Co.Ltd), Sparse-dense wave,20Hz. Stop turning up the current intensity when patients could not stand. 5 times for the first two weeks and 3 times for the last two weeks, 30 min/time.The non-point group take the place 2 cun far from BL33 on the outside horizontally as the non-point and the manipulation methods are the same with those of the point group.
  Other Names: acupuncture; electroacupuncture

SUMMARY:
To evaluate efficacy of BL33 for mild and moderate benign prostatic hyperplasia(BPH).There are trials showing that electroacupuncture on BL33 for mild and moderate BPH is more effective than terazosin. It could reduce the International Prostate Syndrome Score (IPSS) by 6.68±2.84(39.79%),lower urinary symptoms bother of score(BS) and bladder residual urine, and increase maximum urinary flow rate.But the efficacy of BL33 has not been studied. The objective of this study is to evaluate efficacy of BL32 for mild and moderate BPH by comparison with non-acupoint group.

DETAILED DESCRIPTION:
efficacy here means specific effect(or active ingredient) of the point BL33.

ELIGIBILITY:
Inclusion Criteria:

* 50-70 years old
* Mild to moderate BPH evaluated by I-PSS
* Patients having urinary dysfunction more than 3 months
* Patients with stable life signs
* no use of α1 receptor blocker, 5α-reductase inhibitor or traditional Chinese medicine for over 1 week
* Volunteer to join this research and sign the written informed consent prior to receiving treatment

Exclusion Criteria:

* Urinary dysfunction caused by gonorrhea or urinary tract infection
* Oliguria and anuria caused by urinary calculi, prostate cancer, bladder tumor and acute/chronic renal failure
* Urinary dysfunction caused by neurogenic bladder, bladder neck fibrotic and urethral stricture
* Failure of invasive therapy for prostatic obstruction
* Injured local organs, muscle and nerve caused by pelvic operation or historical trauma
* Upper urinary obstruction and hydrocele combined with damaged renal function due to BPH diagnosed by B-ultrasound
* Patients who can't stick to treatment because of economic reason, far distance between home and the hospital or difficult walking etc.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Study Director — Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences
Locations (1):
- Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Wang Y, Liu B, Yu J, Wu J, Wang J, Liu Z. Electroacupuncture for moderate and severe benign prostatic hyperplasia: a randomized controlled trial. PLoS One. 2013 Apr 12;8(4):e59449. doi: 10.1371/journal.pone.0059449. Print 2013. PMID 23593139
- [Derived] Wang Y, Liu Z, Yu J, Ding Y, Liu X. Efficacy of electroacupuncture at Zhongliao point (BL33) for mild and moderate benign prostatic hyperplasia: study protocol for a randomized controlled trial. Trials. 2011 Sep 26;12:211. doi: 10.1186/1745-6215-12-211. PMID 21943105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited patients from BPH clinic by newspaper advertisements and notices at clinic site.192 participants entered the study and 92 of them were excluded.It is supposed that patients with IPSS less than 20 would be included.But few mild BPH patients came for the study.The including criteria were changed and patients with IPSS≥8 were included.
Pre-assignment Details: Diagnosis and assessment were made by an independent urologist who was uninvolved in the treatment process.Baseline assessments included international prostate symptom score (IPSS), postvoid residual urine (PVR) and maximum urinary flow rate (Qmax).
Groups:
- Acupoint: Needle on bilateral BL33 60-80 mm with a 45°angle.A feeling of soreness and distension will be felt when needling into the 3rd posterior sacral foramina(S3).Needle with a 100-125 mm long needle without lifting, thrusting or rotating.An electric stimulator is put on.G6805-2 electric stimulator (produced by Shanghai Huayi Medical Instrument Co.Ltd), Sparse-dense wave,20Hz. Stop turning up the current intensity when patients could not stand. 5 times for the first two weeks and 3 times for the last two weeks, 30 min/time.
  BL33 is an acupuncture point in the Bladder Meridian.Cun is the unit of measurement used in acupuncture, and 1 cun is defined as the distance across the uppermost joint of the thumb of the person being treated.
- Non-acupoint: Take the place 2 cun far from BL33 on the outside horizontally as the non-point. Needle on the non-point for 60-80mm with a 45°angle. A feeling of soreness and distension will be felt .Needle with a 100-125mm long needle without lifting, thrusting or rotating.Sparse-dense wave,20Hz. Stop turning up the current intensity when patients could not stand. 5 times for the first two weeks and 3 times for the last two weeks, 30 min/time.
  BL33 is an acupuncture point in the Bladder Meridian.Cun is the unit of measurement used in acupuncture, and 1 cun is defined as the distance across the uppermost joint of the thumb of the person being treated.
Period: Overall Study
Arm/Group | Acupoint | Non-acupoint
Started | 50 | 50
Treatment Completed | 45 | 42
Completed | 41 | 36
Not Completed | 9 | 14
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupoint | Non-acupoint | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 23 | 47
  >=65 years | 26 | 27 | 53
Age Continuous [Mean (Standard Deviation); unit: years] | 64.8 (7.05) | 65.9 (6.74) | 65.37 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 50 | 100
Region of Enrollment [Number; unit: participants]
  China | 50 | 50 | 100
International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: units on a scale] — Score range:0-35(0 is best，35 is worst, ordinal)
  units on a scale | 20.10 (6.52) | 18.76 (6.06) | 19.43 (6.30)
bladder residual urine [Median (Full Range); unit: ml] | 20 [0 to 128] | 16 [0 to 128] | 20 [0 to 128]
maximum urinary flow rate (Qmax) [Mean (Standard Deviation); unit: ml/s] | 13.04 (6.73) | 15.93 (7.33) | 14.51 (7.15)

OUTCOME MEASURES:

1. Primary Outcome: Change of IPSS at the 6th Week Compared With Baseline(Intention to Treat)
Description: International Prostate Symptom Score (IPSS) Range:0-35(0 is best，35 is worst, ordinal),6 week mean minus baseline mean.And analysis for this outcome measure is based on ITT population.
Time Frame: baseline and the 6th week
Population: The data analysis of the primary outcome was based on the ITT population(data of all participants who are randomized will be analyzed).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupoint | Non-acupoint
Number analyzed (Participants) | 50 | 50
units on a scale | 7.26 (5.12) | 2.34 (4.85)
Statistical Analysis 1: Comparison: Acupoint vs Non-acupoint; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Difference (Net) = 4.51, 95% CI 2-sided [2.67 to 6.36], Standard Error of Mean 0.93

2. Secondary Outcome: Change of Bladder Residual Urine at the 6th Week
Description: Bladder residual urine was used to assess the bladder function, 6 week mean minus baseline mean
Time Frame: baseline and the 6th week
Population: The data analysis of the secondary outcome was based on the ITT population.
Measure: Median (Full Range); unit: ml
Arm/Group | Acupoint | Non-acupoint
Number analyzed (Participants) | 50 | 50
ml | 0 [-172 to 84] | 0 [-120 to 80]
Statistical Analysis 1: Comparison: Acupoint vs Non-acupoint; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 3.34, 95% CI 2-sided [-9.76 to 16.44], Standard Error of Mean 6.60

3. Secondary Outcome: Change of Maximum Urinary Flow Rate(Qmax)at the 6th Week
Description: Maximum urinary flow rate was used to assess the bladder function, 6 week mean minus baseline mean
Time Frame: baseline and the 6th week
Population: The data analysis of the secondary outcome was based on the ITT population.
Measure: Mean (Standard Deviation); unit: ml/second
Arm/Group | Acupoint | Non-acupoint
Number analyzed (Participants) | 50 | 50
ml/second | 0.36 (4.51) | 0.98 (4.05)
Statistical Analysis 1: Comparison: Acupoint vs Non-acupoint; Test type: Superiority or Other; p > 0.05, ANCOVA; Mean Difference (Net) = 0.184, 95% CI 2-sided [-1.41 to 1.78], Standard Error of Mean 0.80

4. Secondary Outcome: Change of International Prostate Symptom Score (IPSS) at the 18th Week
Description: International Prostate Symptom Score (IPSS) Range:0-35(0 is best，35 is worst, ordinal),18 week mean minus baseline mean.
Time Frame: baseline and the 18th week
Population: The data analysis of the secondary outcome was based on the ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupoint | Non-acupoint
Number analyzed (Participants) | 50 | 50
units on a scale | 5.48 (5.16) | 1.8 (5.06)
Statistical Analysis 1: Comparison: Acupoint vs Non-acupoint; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Difference (Net) = 3.2, 95% CI 2-sided [1.36 to 5.05], Standard Error of Mean 0.93

5. Primary Outcome: Change of International Prostate Symptom Score(IPSS) at the 6th Week Compared With Baseline(Per-protocol).
Description: International Prostate Symptom Score (IPSS) Range:0-35(0 is best，35 is worst, ordinal),6 week mean minus baseline mean. And analysis for this outcome measure is based on per-protocol population.
Time Frame: baseline and the 6th week
Population: The data analysis of the primary outcome is also based on per-protocol (PP) population as a supportive analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupoint | Non-acupoint
Number analyzed (Participants) | 45 | 42
units on a scale | 7.24 (5.23) | 2.79 (5.17)
Statistical Analysis 1: Comparison: Acupoint vs Non-acupoint; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Difference (Net) = 4.12, 95% CI 2-sided [2.07 to 6.18], Standard Error of Mean 1.03

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Acupoint | Non-acupoint
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 2/50
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Acupoint (N=50) | Non-acupoint (N=50)
ecchymoma (Skin and subcutaneous tissue disorders) | 0/2 (0) | 2/2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes